CLINICAL TRIAL: NCT06512337
Title: A Prospective Observational Study to Evaluate the Effectiveness of Deucravacitinib in Patients With Moderate Plaque Psoriasis in Real-World Settings in China (ADMIRE)
Brief Title: A Observational Study to Evaluate Deucravacitinib in Patients With Moderate Plaque Psoriasis in China
Acronym: ADMIRE
Status: Recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM011-1180
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Plaque Psoriasis
Keywords: Plaque psoriasis
MeSH Terms: interventions — deucravacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants treated with deucravacitinib: Adults with moderate plaque psoriasis who are newly initiating deucravacitinib according to the product label
  Interventions: Drug: Deucravacitinib

INTERVENTIONS:
Drug: Deucravacitinib — As per product label

SUMMARY:
The purpose of this study is to collect and evaluate real-world data on the effectiveness of deucravacitinib treatment in adults with moderate plaque psoriasis in China.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 years or older
* Physician-reported (dermatologist) diagnosis of moderate plaque psoriasis with Body Surface Area ≥ 3% and < 10%
* Participant newly initiated deucravacitinib according to the label
* Provided written informed consent to participate in the study

Exclusion Criteria:

* Participating in or planning to participate in an interventional clinical trial
* Concomitant use of other systemic treatments for psoriasis at baseline
* Prior treatment of deucravacitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants aged ≥ 18 years who have been diagnosed with moderate plaque psoriasis who are starting deucravacitinib treatment in China
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving Static Physician's Global Assessment (sPGA) 0/1 score | Week 16
Participant psoriasis Body Surface Area (BSA) involvement | Week 16
Number of participants achieving absolute Psoriasis Area and Severity Index (PASI) score ≤ 3 | Week 16

SECONDARY OUTCOMES:
Number of participants achieving Psoriasis Area and Severity Index (PASI) 75 response and PASI 90 response | Baseline and Weeks 4, 12, 24, 36, and 52
Number of participants achieving absolute Psoriasis Area and Severity Index (PASI) score ≤1, ≤2, ≤3, and ≤5 | Baseline and Weeks 4, 12, 24, 36, and 52
Participants change in Participant Absolute Psoriasis Area and Severity Index (PASI) score from baseline | Weeks 4, 12, 16, 24, 36, and 52
Number of participants achieving psoriasis Body Surface Area (BSA) involvement of ≤1% and ≤3% | Baseline and Weeks 4, 12, 16, 24, 36, and 52
Change in Body Surface Area (BSA) involvement from baseline to follow-up | Weeks 4, 12, 24, 36, and 52
Static Physician's Global Assessment (sPGA) 0/1 response at follow-up | Weeks 4, 12, 24, 36, and 52
Participants change in Static Physician's Global Assessment (sPGA) score from baseline | Baseline and Weeks 4, 12, 16, 24, 36, and 52
Number of participants achieving a Dermatology Life Quality Index (DLQI) 0/1 score | Baseline and Weeks 4, 12, 16, 24, 36, and 52
Number of participants achieving a Dermatology Life Quality Index (DLQI) ≤ 3 score | Baseline and Weeks 4, 12, 16, 24, 36, and 52
Change in participant Dermatology Life Quality Index (DLQI) score from baseline | Baseline and Weeks 4, 12, 16, 24, 36, and 52

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- China (5):
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Affiliated Hospital of Hebei University of Engineering, Handan, Hebei
  - DaLian Dermatosis Hospital, Dalian, Liaoning
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts